CLINICAL TRIAL: NCT06012721
Title: A Phase 1, Randomized, Open-Label, Crossover Study Evaluating the Effect of Food on the Pharmacokinetics of ORIC-114 Tablet Formulation in Healthy Subjects
Brief Title: Effect of Food on the Pharmacokinetics of ORIC-114
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ORIC Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ORIC-114-03
Record Dates: First submitted 2023-08-17; First posted 2023-08-25 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Food Effect in Healthy Participants
Keywords: Food effect; ORIC-114

STUDY DESIGN:
Intervention Model Description: Randomized, 2-part, 2-sequence, 2-period, open-label, crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part 1 Treatment A (Experimental): 30 mg ORIC-114 (3 x 10 mg tablets) administered at Hour 0 on Day 1 under fasting conditions.
  Interventions: Drug: ORIC-114
- Part 1 Treatment B (Experimental): 30 mg ORIC 114 (3 x 10 mg tablets) administered at Hour 0 on Day 1, 30 minutes after the start of a meal.
  Interventions: Drug: ORIC-114
- Part 2 Treatment A (Experimental): xx mg ORIC-114 (n x 10 mg tablets) administered at Hour 0 on Day 1 under fasting conditions.
  Interventions: Drug: ORIC-114
- Part 2 Treatment B (Experimental): xx mg ORIC 114 (n x 10 mg tablets) administered at Hour 0 on Day 1, 30 minutes after the start of a meal.
  Interventions: Drug: ORIC-114

INTERVENTIONS:
Drug: ORIC-114 — Food effect healthy subjects

SUMMARY:
A randomized, 2-part, 2-sequence, 2-period, open-label, crossover study evaluating the effect of food on the pharmacokinetics (PK) of ORIC-114 tablet formulation in healthy adult subjects.

DETAILED DESCRIPTION:
The study will be performed in two parts. Part 1 will assess the effect of food at a lower dose of ORIC-114 to first ascertain the degree of food effect (if any) on ORIC-114 exposure as a way to ensure the safety of the participating subjects. Part 2 will further assess the food effect at a higher dose of ORIC-114.

If the preliminary Part 1 results clearly show no food effect, Part 2 may not need to be conducted upon assessment by the Sponsor.

If Part 2 is conducted, the dose of ORIC-114 will be selected within the anticipated efficacious clinical dose range based on results from Part 1.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male or female (of nonchildbearing potential only), 18-55 years of age
2. Continuous nonsmoker who has not used nicotine and tobacco containing products for at least 30 days
3. Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2
4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, and ECGs, as deemed by the PI or designee
5. Able to swallow multiple tablets.

Exclusion Criteria:

1. Mentally or legally incapacitated or has significant emotional problems
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
3. History or presence of alcohol or drug abuse within the past 2 years prior to the first dosing.
4. History or presence of clinically significant GI disorder (
5. Female subjects of childbearing potential.
6. Positive urine drug screen or alcohol breath test results
7. Positive results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV)
8. Lactose intolerant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | 14 days
  To evaluate the effect of food on the single dose PK of ORIC-114 tablet formulation
Time of maximum observed concentration (Tmax) | 14 days
  Food Effect: PK of ORIC-114 tablet
Area under the curve (AUC) | 14 days
  Food Effect: PK of ORIC-114 tablet
Apparent plasma terminal elimination half-life (t1/2) | 14 days
  Food Effect: PK of ORIC-114 tablet

SECONDARY OUTCOMES:
Number of subjects with Treatment Emergent Adverse Effect | 30 days
  Assessed by NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Pratik S Multani, MD, MS, Study Director — ORIC Pharmaceuticals
Locations (2):
- Australia (2):
  - Nucleus Network Pty Ltd., 235 Ryrie St, Geelong, Victoria
  - Nucleus Network Pty Ltd., Level 5, Burnet Tower, 89 Commercial Rd, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No